CLINICAL TRIAL: NCT05542901
Title: The Comparison of Joint Position Sense in Diabetic and Traumatic Transtibial Amputees and The Investigation of The Relationship Between Compliance With a Prosthesis, Balance, and Functional Performance With Joint Position Sense
Brief Title: Comparison of Joint Position Sense in Diabetic and Traumatic Transtibial Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Melek Merve ERDEM, Research Assistant, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: GO 21/1101
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Diabetic Polyneuropathy; Amputation
Keywords: Diabetic Polyneuropathy; Lower Extremity Amputation; Joint Position Sense; Compliance With The Prosthesis; Balance; Functional Performance
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic Group (DG) (Other): Examine the effect of joint position sense on compliance with the prosthesis, balance and functional performance in individuals with lower extremity amputation due to diabetic polyneuropathy.
  Interventions: Diagnostic Test: Joint Position Sense Analysis
- Traumatic Group (TG) (Other): Examine the effect of joint position sense on compliance with the prosthesis, balance and functional performance in individuals with lower extremity amputation due to traumatic causes.
  Interventions: Diagnostic Test: Joint Position Sense Analysis

INTERVENTIONS:
Diagnostic Test: Joint Position Sense Analysis — The Xsens DOT Motion Capture System will be used to analyze joint position sense.

SUMMARY:
This study evaluated the effect of joint position sense on compliance with the prosthesis, balance and functional performance in individuals with lower extremity amputation due to diabetic polyneuropathy. Study group consisted of 16 subjects with unilateral transtibial amputation due to diabetic polyneuropathy and control group consisted of 16 subjects with unilateral transtibial amputation due to traumatic reasons.

DETAILED DESCRIPTION:
Proprioception is defined as the ability to distinguish the position of various body parts relative to each other and the ground through the sensory system (kinesthesia) and to perceive the forces acting on these body parts. Proprioception is a function that takes place mainly on a subconscious level. Information about the external environment we live in is obtained from the combination of nerve terminals in muscles and tendons, fibrous capsules around joints, vestibular and visual systems. The proprioceptive information obtained about the external environment through the peripheral nervous system is transferred to the central nervous system. The integration of these data collected from different sensory receptors is performed, and appropriate motor responses are initiated to ensure postural balance. Sensory loss due to pain, fatigue, effusion, trauma, or various neurological, musculoskeletal disorders and metabolic diseases such as diabetes often causes a decrease in proprioceptive sensation in these case groups. Peripheral nerve damage due to diabetic polyneuropathy (DPN), varies depending on the type of nerve fiber affected. As a result of damage to unmyelinated and small myelinated nerve fibers, light touch, pain and temperature senses are impaired while vibration and proprioception senses are decreased as a result of damage to large myelinated nerve fibers. Recent studies have shown that individuals with DPN are more likely to apply to the emergency department due to complications from fall accidents because they experience balance loss during activities of daily living compared to healthy non-diabetic individuals. Furthermore, foot biomechanics, which deteriorates owing to the loss of the normal neural feedback system caused by DPN, causes foot ulcerations by creating aberrant pressure distribution in the foot. In these people, non-healing lower limb ulcers account for 85% of planned lower extremity amputations. Due to the predicted loss of soft tissue, bone, and sensory receptors in the amputated limb following a prior lower extremity amputation, which results in musculoskeletal system degradation and destruction of the mechanoreceptors innervating these tissues, the way these individuals experience their surroundings changes and differentiates them from individuals who have been amputated due to traumatic causes. Diabetic amputees are unable to utilize their prostheses functionally following amputation due to their physical problems, which results in the majority of patients discontinuing usage of prosthesis. Although the number of test batteries developed to assess proprioceptive sense and the effectiveness of rehabilitation protocols used to assess proprioceptive sense in individuals with musculoskeletal disorders such as amputation is insufficient in the literature, it is believed that the existing batteries do not adequately assess proprioceptive sense. Additionally, no study has been conducted to determine the extent to which these patients' proprioceptive sensibility is altered following lower limb amputation due to DPN. For this reason, the study was planned to examine the effect of joint position sense on compliance with the prosthesis, balance and functional performance in individuals with lower extremity amputation due to DPN.

ELIGIBILITY:
Inclusion Criteria:

Diabetic Group (DG):

1. Those who had unilateral transtibial amputation due to DPN
2. Between the ages of 40-65
3. Completed rehabilitation with prosthesis
4. Using prosthesis for at least 1 year
5. With standard size stump length
6. Without phantom sensation and pain
7. Able to walk at least 10 m independently
8. Gross lower extremity muscle strength at least moderate
9. No cognitive and mental problems
10. Diabetic nephropathy, retinopathy, ulceration etc. without secondary complications
11. Those who voluntarily agreed to participate in the research
12. Not included in any other concurrent study

Traumatic Group (TG):

1. Those who had trauma-induced unilateral transtibial amputation
2. Between the ages of 40-65
3. Completed rehabilitation with prosthesis
4. Using prosthesis for at least 1 year
5. With standard size stump length
6. Without phantom sensation and pain
7. Able to walk at least 10 m independently
8. Gross lower extremity muscle strength is at least moderate
9. Absence of cognitive and mental problems
10. Those who voluntarily agreed to participate in the research
11. Not included in any other concurrent study

Exclusion Criteria:

For all groups;

1. Having osteoarticular deformity in the knee joint
2. Having an orthopedic or neurological disease other than the cause of amputation
3. Significant and irreversible visual deficit
4. Body mass index (BMI)>30 kg/m²
5. Having a disability that makes it hard to complete any of the tests
6. Individuals with a history of cancer and receiving chemotherapy

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Joint Position Sense | 1 week
  The Xsens DOT Motion Capture System will be used in the evaluation of knee joint proprioception. . Before starting the measurement, the sensors are properly attached to the patient. The sense of proprioception of the knee joint will be evaluated bilaterally with weightless (NWB) using the method. The NWB assessment will be performed with and without prosthesis while the person is in a sitting position with their legs fully supported. The person's eyes will be covered with a band aid to avoid any visual cues. The knee joint in extension position will be slowly brought to the target angle value of 30° and 60° flexion position by the physiotherapist and waited for 4 seconds. After 3 consecutive attempts, the participant will be asked to actively perform the flexion movement whose angle is determined using the same limb. There will be 2 minute rest breaks between measurements. The difference between the target angle and the measured angle is recorded as the margin of error.

SECONDARY OUTCOMES:
The Limits of Stability | 1 week
  The limits of stability were used to evaluate static balance. Limits of stability is the greatest distance in any direction a person can lean away from a midline vertical position without falling, stepping, or reaching for support. Participants were assessed with a force platform (Model BP 5050; Bertec Corporation, Columbus, Ohio) in terms of support surfaces on limits of stability (LoS) in the right, left, front and back directions when the eyes were open on the hard floor with the Bertec Balance System on their preferred support surface width.
Postural Sway | 1 week
  Postural sways were used to evaluate dynamic balance. Postural sway, in terms of human sense of balance, refers to horizontal movement around the center of gravity. Postural sway was measured while quiet standing with open/closed eyes on a hard/soft floor using the Bertec Balance System at their preferred support surface width.
Functional Capacity | 1 week
  2 Minute Walk test was used to evaluate the functional capacity. The test was performed in a corridor on a flat hard surface of 30 m in length in a straight line. Before the examination, the patient rested for 10 min in a sitting position. It is calculated by measuring the distance that the person walks at the end of this period by asking the person to walk for 2 minutes along a 30 m corridor. In cases of chest pain, dyspnea, leg cramps, excessive fatigue, sweating and wilting, the test should be terminated immediately. At one-minute intervals during the test, the participant received information about the time remaining until the end of the test.

CONTACTS AND LOCATIONS:
Overall Officials: Melek M. ERDEM, PT, M.Sc., Principal Investigator — Tayyip Erdogan University Training and Research Hospital; Semra TOPUZ, PT, Prof., Study Director — Hacettepe University; Ali I. YALCIN, PT, Ph.D., Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available within 3 months with completion of the result report.
Access Criteria: Requestors will be required to sign a Data Access Agreement.
URL: https://orcid.org/0000-0003-4073-3084

REFERENCES:
- [Background] Fontes Filho CHDS, Laett CT, Gavilao UF, Campos JC Jr, Alexandre DJA, Cossich VRA, Sousa EB. Bodyweight distribution between limbs, muscle strength, and proprioception in traumatic transtibial amputees: a cross-sectional study. Clinics (Sao Paulo). 2021 Apr 26;76:e2486. doi: 10.6061/clinics/2021/e2486. eCollection 2021. PMID 33909824